CLINICAL TRIAL: NCT03874936
Title: The Effect of Perioperative Dexamethasone Administration on Postoperative Pain in Patients Undergoing Periacetabular Osteotomy: A Randomised Double-blind, Placebo-controlled Trial
Brief Title: The Effect of Perioperative Dexamethasone Administration on Postoperative Pain in Patients Undergoing Periacetabular Osteotomy.
Acronym: PAODEX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Viktoria Lindberg-Larsen, MD, PhD, principal investigator and sponsor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SO_SH_01_2019; 2019_000402_30 (EudraCT Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Dexamethasone; Hip Dysplasia; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: postoperative pain; dexamethasone; pain management
MeSH Terms: conditions — Hip Dislocation; Pain, Postoperative; Postoperative Nausea and Vomiting; Agnosia | interventions — Dexamethasone; Solutions; Injections; Absorptiometry, Photon; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A; Dexamethasone twice (Experimental): 24mg intravenous Dexamethasone (Dexavital®, Vital Pharma) 4mg/ml just before the operation and repeated after 24 hours.
  Interventions: Drug: Dexamethasone 24mg Solution for Injection
- B; Dexamethasone once (Experimental): 24mg intravenous Dexamethasone just before the operation and placebo which is 6ml of isotonic sodium chloride (9mg/ml, 'normal' saline) after 24 hours
  Interventions: Drug: Dexamethasone 24mg Solution for Injection; Drug: Saline Solution for Injection
- C; Placebo twice (Placebo Comparator): placebo intravenous just before the operation and repeated after 24 hours
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Dexamethasone 24mg Solution for Injection — Administrated i.v.
  Other Names: Dexa
  Arms: A; Dexamethasone twice; B; Dexamethasone once
Drug: Saline Solution for Injection — administrated i.v.
  Other Names: Saline
  Arms: B; Dexamethasone once; C; Placebo twice

SUMMARY:
This is an investigator-initiated, Danish mono-center, randomized, placebo-controlled, parallel group, double-blind, superiority trial of dexamethasone on postoperative pain management on patients undergoing operation for hip dysplasia with the periacetabular osteotomy procedure (PAO). 90 adults undergoing PAO will be enrolled.

The primary outcome is to compare the effect of dexamethasone relative to placebo on cumulated postoperative morphine consumption at 48 hours.

Key secondary outcomes include comparing the effect of repeated doses of dexamethasone relative to a single dose on cumulated postoperative morphine consumption at 48 hours, and to determine if dexamethasone is superior to placebo for: Perception of pain intensity, prevalence and degree of postoperative nausea and vomiting, and patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PAO due to symptomatic hip dysplasia (CE<25grader) or retroverted acetabulum (crossover and posterior wall sign)
* ≥ 18 years
* Females if fertile: Verified negative human chorionic gonadotropin (HCG), usage of safe contraceptives or surgical sterilisation.
* Patients who give their written informed consent to participating in the trial, after having fully understood the content of the protocol and restrictions.

Exclusion Criteria:

* Patients who cannot speak or understand Danish
* Allergy or contraindications to trial medication
* Spinal anaesthesia
* Second intervention carried out simultaneously (e.g. femur osteotomy)
* Patients with daily opioid consumption prior to surgery (tramadol and codeine accepted)
* Drug, medical abuse or weekly alcohol consumption beyond ≥7 (female) and ≥14 (men) units, respectively.
* Mental disability, anxiety disorder (active psychiatric disorder or consumption of tricyclic antidepressants)
* Diabetes diagnosed prior to inclusion
* Immune suppression therapy (e.g. systemic glucocorticoids)
* Kidney impairment (eGFR < 50ml/min) or liver disease (≥Child Pugh B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulated postoperative morphine consumption in milligrams after 48 hours. | 0-48 hours postoperatively
  Morphine administered both as patient-controlled analgesia (PCA) i.v. morphine and any other supplemental morphine administered postoperatively. Consumption in mg.

SECONDARY OUTCOMES:
Postoperative pain intensity after 48 hours. | 24, 48 hours postoperatively
  Pain is evaluated at rest and under the timed-up-and-go (TUG) procedure. Pain intensity is assessed using the visual analogue scale (VAS) (0-100mm).
Cumulated postoperative morphine consumption from 48 hours until day 14 post operation | 48 hours - day 14 postoperatively
  Morphine consumption in milligrams after the operation.
Postoperative nausea and vomiting | 24 and 48 hours postoperatively
  Nausea and vomiting are evaluated using a 4 point scale: none, mild, moderate, severe
Antiemetic consumption | 0-48 hours postoperatively
  Evaluation of cumulated antiemetic consumption in mg and drug will be assessed.
Sleep | 0-7 days postoperatively
  Sleep quality will be assessed using the VAS scale (0-100)
Timed up and go test | 24, 48 hours postoperatively
  Is assessed from; the time that the participant takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Serious adverse events (SAE) | 0-8 weeks after operation
  SAE's including wound infection treated with antibiotics or revision. Patients will be asked for SAE during the intervention period, at a follow-up visit 8 weeks the operation. This will be supplemented with a look up for prescriptions.

OTHER OUTCOMES:
Cumulated postoperative morphine consumption in milligrams after 24hours. | 0-24 hours postoperatively
  Morphine administered both as patient-controlled analgesia (PCA) i.v. morphine and any other supplemental morphine administered postoperatively. Consumption in mg.
Cumulated antiemetic consumption | 0-24 hours postoperatively
  antiemetic consumption in mg and drug will be assessed after 24hrs.
Fasting blood glucose | 0 hours, 6 hours, 24 hours, 48 hours (72 hours)
  assessment of fasting blood glucose in mg/mL
C-reactive protein (CRP) | 0, 6, 24, 48 hours (72 hours) postoperatively
  blood sample to evaluate the influence of dexamethasone on the postoperative inflammation development.
Leucocytes | 0, 6, 24, 48 hours (72 hours) postoperatively
  blood sample to evaluate the influence of dexamethasone on the postoperative inflammation development.
Cytokines | 0, 6, 24, 48 hours (72 hours) postoperatively
  evaluate the decrease of cytokines concentration (Interleukin (IL)-2, IL-6, IL-10, tumor necrosis factor (TNF) and pentraxin 3 (PTX3) as markers of response during treatment with Dexamethasone
Patient reported outcome measure, quality of life | 3, 6, 12 months postoperatively
  Based on the questionnaire: EuroQol - 5 Dimensions (EQ-5D) after 3 and 6 months and 1 year follow up.
Patient reported outcome measures, health | 3, 6, 12 months postoperatively
  Patient evaluated health based on the questionnaire: University of California, Los Angeles (UCLA) after 3 and 6 months and 1 year follow up.
Patient reported outcome measures, the Oxford Hip questionnaire | 3, 6, 12 months postoperatively
  Patient evaluated activity and pain, based on the questionnaire: Oxford Hip after 3 and 6 months and 1 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, PhD, Study Chair — Dept. of Anesthesiology and Intensive Care Medicine, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindberg-Larsen V, Lindberg-Larsen M, Ovesen O, Zwisler ST, Lindholm P, Hebsgaard S, Christensen R, Overgaard S. Effect of high-dose dexamethasone on morphine use after periacetabular osteotomy for hip dysplasia: a randomized double-blind placebo-controlled single center trial. Acta Orthop. 2025 Jun 1;96:413-420. doi: 10.2340/17453674.2025.43903. PMID 40460271

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT03874936/SAP_000.pdf